CLINICAL TRIAL: NCT03913793
Title: Impact of Peripheral Neuropathy in Type-II Diabetes Mellitus on Outcome Measures of Weight-Bearing Aerobic Training in Post-Myocardial Infarction Patients.
Brief Title: Aerobic Training in Post-MI Patients With DPN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yousra Hisham Abdel Fattah (Other)
Collaborators: Diaa Mohamed Mohasseb (Unknown); Mahmoud Mohamed Hassanein (Unknown); Gihan Younis El-tantawi (Unknown); Aya Hanafy Ibrahiem (Unknown)
Responsible Party: Sponsor-Investigator, Yousra Hisham Abdel Fattah, Principle investigator, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0104363
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Myocardial Infarction; Diabetes Mellitus, Type 2; Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Myocardial Infarction; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuropathy group (Active Comparator): post-myocardial infarction patients with type-II diabetes mellitus enrolled in the study within 1-6 months of myocardial infarction with peripheral neuropathy , enrolled into exercise program From those referred for cardiac rehabilitation in the cardiac rehabilitation unit, Alexandria Teaching Hospital
  Interventions: Other: Exercise based-cardiac rehabilitation (EB-CR) program
- Non-Neuropathy group (Active Comparator): post-myocardial infarction patients with type-II diabetes mellitus enrolled in the study within 1-6 months of myocardial infarction without peripheral neuropathy , enrolled into exercise program From those referred for cardiac rehabilitation in the cardiac rehabilitation unit, Alexandria Teaching Hospital
  Interventions: Other: Exercise based-cardiac rehabilitation (EB-CR) program
- Control group (No Intervention): post-myocardial infarction patients with type-II diabetes mellitus enrolled in the study within 1-6 months of myocardial infarction, not enrolled into exercise program.

INTERVENTIONS:
Other: Exercise based-cardiac rehabilitation (EB-CR) program — The exercise group underwent an outpatient EB-CR program (phase II) according to the American College of Sports Medicine guidelines for exercise prescription for cardiac patients.[19] Sessions were 3 days/week for 8 weeks. The program included: (1) Warm up (10 minutes): stretching exercises. (2) Aerobic exercise training using treadmill (30 - 60 minutes/session): with target heart rate (HR) at 45 - 75% of HR reserve. The maximal HR (HR max) was derived from that obtained during exercise stress test (EST). Patients who had ischemic/arrhythmic manifestations during EST, exercise intensity was prescribed at a HR below the ischemic threshold (10 beats below). (3) Cool down (10 minutes): light intensity treadmill walking. Supervision was provided according to the risk status of each patient that was determined according to the American Association of cardiovascular and Pulmonary Rehabilitation criteria for risk stratification.
  Arms: Neuropathy group; Non-Neuropathy group

SUMMARY:
Cardiac rehabilitation (CR) is categorized by the American College of Cardiology "class IA recommendation" in the management of patients with cardiovascular disease (CVD) including post-myocardial infarction (MI) patients, who have reduced functional capacity and impaired quality of life. Studies have reported that post-MI patients enrolled in exercise-based CR (EB-CR) show improved functional capacity, significant decrease risk of re-infarction, and 25% reduction in mortality. Aim: To define the effect of diabetic peripheral neuropathy (DPN) on the outcome measures of exercise based-cardiac rehabilitation (EB-CR) program in post-myocardial infarction (MI) patients with type-II diabetes mellitus (DM).

Methods: Thirty-seven post-MI patients with type-II DM were enrolled in the study within 1-6 months of MI from those referred for cardiac rehabilitation in the cardiac rehabilitation unit, Alexandria Teaching Hospital. Seven patients were lost. Fifteen patients attended 8 weeks of aerobic training program (exercise group; 12 men and 3 women) while 15 patients did not (control group; 11 men and 4 women). The exercise group was assessed for the presence of peripheral neuropathy and patients were accordingly subdivided into those with DPN "group A" and those without "group B". All groups were evaluated at baseline and at the end of the study. Evaluation included Duke Activity Status Index (DASI) questionnaire, 6-minute walk test, and symptom-limited treadmill exercise stress test (EST).

Outcome measures included: DASI score; 6-minute walk test distance (6MWD); and heart rate (HR), blood pressure (BP), rate pressure product (RPP), and functional capacity in metabolic equivalents (METs) measured during EST.

DETAILED DESCRIPTION:
The study population included post-MI patients with type-II DM within 1 to 6 months from onset of MI from those referred for cardiac rehabilitation in the cardiac rehabilitation unit, Alexandria Teaching Hospital. Patients were diagnosed as having MI according to the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of MI and DM according to the 2016 American Diabetes Association guidelines.

All patients were assessed by a cardiologist by clinical examination, electrocardiogram and echocardiography. Patients were excluded if they had any contraindication to exercise stress test (EST) or CR,systemic illness other than DM or hypertension, neurological disorders other than DPN, or had loss of protective sensation (anesthesia) and/or ulcerations in the lower limbs.

All patients were informed about the nature of the study and an informed consent was obtained from all of them. The protocol was approved by the ethics committee.

Patients were divided into 2 groups; those enrolled in EB-CR program "exercise group" and those not enrolled in EB-CR program "control group".

Baseline evaluation for both groups included: demographic data collection, history taking, clinical examination, electrophysiological studies to confirm the presence or absence of neuropathy (sural sensory, posterior tibial and deep peroneal motor conduction studies), total neuropathy score to assess the clinical severity of DPN, Duke Activity Status Index questionnaire (DASI) to assess patients' physical activity level, Six-Minute Walk Test, and symptom-limited treadmill EST using Bruce protocol. All patients were on their regular medications including B-blockers during the EST.

The exercise group underwent an outpatient EB-CR program (phase II) according to the American College of Sports Medicine guidelines for exercise prescription for cardiac patients.Sessions were 3 days/week for 8 weeks. The program included: Warm up (10 minutes): stretching exercises. Aerobic exercise training using treadmill (30 - 60 minutes/session): with target heart rate (HR) at 45 - 75% of HR reserve. The maximal HR (HR max) was derived from that obtained during EST. Patients who had ischemic/arrhythmic manifestations during EST, exercise intensity was prescribed at a HR below the ischemic threshold (10 beats below). Cool down (10 minutes): light intensity treadmill walking. Supervision was provided according to the risk status of each patient that was determined according to the American Association of cardiovascular and Pulmonary Rehabilitation criteria for risk stratification. Controls were advised to maintain their medications and regular activities of daily living.

The follow-up evaluation included: DASI, Six Minute Walk Test and symptom limited EST. The Outcome measures were DASI score, Six-minute walk test distance (6MWD), functional capacity in metabolic equivalents (METs), HR, blood pressure (BP) and rate pressure product (RPP) at a given workload.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as having MI according to the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of MI
* DM according to the 2016 American Diabetes Association guidelines

Exclusion Criteria:

* contraindication to exercise stress test (EST)
* contraindication to cardiac rehabilitation,
* systemic illness other than DM or hypertension,
* neurological disorders other than DPN,
* had loss of protective sensation (anesthesia)
* had ulcerations in the lower limbs.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Duke Activity Status Index (DASI) questionnaire | 8 weeks
  12 questions of self-administered questionnaire that measures a patient's functional capacity, The index included questions about activities of daily living as personal care, house hold activities and recreational activities. It also correlated activities with peak oxygen uptake.
  Maximum value 58.2 and Minimum value 0, higher values indicate better functional capacity.
  Estimated peak oxygen uptake in mL/min = (0.43 * (duke activity status index) + 9.6
heart rate (HR) | 8 weeks
  number of heart beats per minute,
blood pressure (BP), | 8 weeks
  systolic and diastolic blood pressure in mmHg
rate pressure product (RPP), | 8 weeks
  is a measure of the stress put on the cardiac muscle based on the number of times it needs to beat per minute (HR) and the arterial blood pressure that it is pumping against
Six minute walk test distance | 8 weeks
  It is used to estimate the functional capacity of the study group. It was done according to the American Thoracic Society (ATS) guidelines for the 6MWT.
  The 6MWT was performed in an indoors flat straight corridor of 30 meters in length. A stopwatch was used to measure the 6 minutes. Patients were instructed that the target of the test was to: WALK AS FAR AS POSSIBLE for 6 minutes, WITHOUT RUNNING OR JOGGING

IPD SHARING:
Plan to Share IPD: No